CLINICAL TRIAL: NCT02474524
Title: Psychosocial Intervention Using Online Resources to Promote Personal Recovery in Users of Specialist Mental Health Services
Brief Title: Self-Management and Recovery Technology Psychosocial Intervention Trial
Acronym: SMARTTherapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Swinburne University of Technology (Other)
Collaborators: The Alfred (Other); St Vincent's Hospital Melbourne (Other); Melbourne Health (Other); Mental Illness Fellowship of Victoria (Unknown); Mind Australia (Other); La Trobe University (Other); Deakin University (Other); Austin Health (Other Government); Neami National (Unknown); Peninsula Health (Other Government); Eastern Health (Other); EACH (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2014/119; MIRF33 (Other Grant/Funding Number: Victorian Department of Health Mental Illness Research Fund)
Record Dates: First submitted 2015-05-24; First posted 2015-06-17 (Estimated); Last update posted 2017-09-15 (Actual); Status verified 2017-09

CONDITIONS: Schizophrenia; Affective Disorders, Psychotic; Psychotic Disorders
Keywords: Psychosis; Schizophrenia; Self-management; Recovery; Tablet computer; Digital health; Internet; Online; Peer support
MeSH Terms: conditions — Schizophrenia; Affective Disorders, Psychotic; Psychotic Disorders | interventions — Play Therapy; Social Work

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Health intervention (Experimental): + treatment as usual
  Interventions: Behavioral: Health intervention
- Social intervention (Active Comparator): + treatment as usual
  Interventions: Behavioral: Social intervention

INTERVENTIONS:
Behavioral: Health intervention — Participants will receive 8 50-minute sessions during a 3 month window with a mental health worker, in addition to their routine care. Sessions will be structured by the worker and participant using a tablet computer to view materials on mental health self-management and personal recovery on a dedicated website for the trial. These will include information, videos, audio and exercises. Online materials make particular use of videos featuring people with lived experience of psychosis discussing how they have dealt with issues in their recovery, and will allow users to post comments on videos and in a forum. Participants may access online materials both during intervention sessions and outside sessions using any Internet-enabled device.
  Arms: Health intervention
Behavioral: Social intervention — Participants will receive 8 50-minute sessions during a 3 month window with a mental health worker in addition to routine care (treatment as usual). The social intervention will utilise a computer tablet (i.e., iPad) servicing online resources to extend a manualised befriending intervention, based upon social interaction, designed to control for therapist contact and computer use. Each session will involve interaction about non-health related topics of interest to the participants, which will be facilitated by use of viewing online material related to these interests on a tablet computer as a prompt to conversation.
  Arms: Social intervention

SUMMARY:
This project is a component of a broader research program referred to as "Self-Management and Recovery Technology (SMART): Use of online technology to promote self-management and recovery in people with psychosis", which has been funded by the Victorian Department of Health Mental Illness Research Fund (MIRF33). The overall research program is examining the therapeutic potential of using online (Internet-based) educational and multimedia resources in mental health services. It involves the development of a website which can be accessed via an internet browser on a desktop computer, tablet computer, or smartphone. It consists of a series of educational modules containing textual information, exercises, audio, and video clips designed to promote self-management and recovery in people with a history of persisting mental illness.

This particular project (SMART-Therapy) involves a randomised controlled trial examining the use of a discrete 8-session psychosocial intervention delivered in addition to routine care which utilises these online materials. The intervention will involve a mental health worker meeting with the participant with a tablet computer (e.g. iPad) on which online materials can be viewed, and used to guide an interaction with the participant.

The randomised controlled trial will include 148 participants, who will be randomised to receive one of two interventions: (a) meeting with a support worker using the SMART website to guide interaction (health intervention), or (b) meeting with a support worker delivering a social interaction-based control condition (social intervention). In each condition, there will be 8 x 50min face-to-face sessions over 3 months. Assessments will be completed pre-randomisation, and at 3, 6 and 9 months.

The primary hypothesis is that participants randomised to the health intervention will show greater improvement in personal recovery than participants randomised to the social intervention, and that these improvements will be maintained at follow-up (6 and 9 months following intake).

ELIGIBILITY:
Inclusion Criteria:

1. diagnosis of a functional psychotic disorder (schizophrenia-related disorder OR bipolar disorder or major depressive disorder with the presence of a severe episode with psychotic features within the past 2 years);
2. sufficient fluency in English to make use of the resources;
3. overall intellectual functioning within normal limits (WTAR estimated IQ>70);

Exclusion criteria (e) change in medication or in-patient admission in the previous 2 months;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2017-06 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
Change in Process of Recovery Questionnaire (QPR) | Baseline, 3, 6 and 9 months
  Assesses personal recovery

SECONDARY OUTCOMES:
Change in Positive and Negative Syndrome Scales (PANSS) | Baseline, 3, 6 and 9 months
  Assesses psychotic symptomatology
Change in Subjective Experience of Psychosis Scale (SEPS) | Baseline, 3, 6 and 9 months
  Assesses subjective impact of psychotic symptoms
Change in Depression Anxiety Stress Scale (DASS-21) | Baseline, 3, 6 and 9 months
  Assesses emotional symptoms
Change in Assessment of Quality of Life 8dimension (AQol8d) | Baseline, 3, 6 and 9 months
  Assesses quality of life
Change in Resource Use Questionnaire | Baseline, 3, 6 and 9 months
  Measure of health service use

OTHER OUTCOMES:
Change in Self-Efficacy for Personal Recovery Scale | Baseline, 3, 6 and 9 months
Change in General Self-Efficacy Scale | Baseline, 3, 6 and 9 months
Change in Schizophrenia Hope Scale | Baseline, 3, 6 and 9 months
Change in UCLA Loneliness Scale | Baseline, 3, 6 and 9 months
Change in Internalised Stigma of Mental Illness Scale | Baseline, 3, 6 and 9 months

CONTACTS AND LOCATIONS:
Overall Officials: Neil Thomas, Principal Investigator — Swinburne University of Technology/Alfred Health
Locations (10):
- Australia (10):
  - EACH, Eastern Melbourne, Victoria
  - Eastern Health, Eastern Melbourne, Victoria
  - Mental Illness Fellowship of Victoria, Fairfield, Victoria
  - St Vincent's Health mental health services, Fitzroy, Victoria
  - Peninsula Health, Frankston, Victoria
  - Austin Health, Heidelberg, Victoria
  - Mind Australia, Heidelberg, Victoria
  - Alfred Health mental health services, Melbourne, Victoria
  - Neami National, Melbourne, Victoria
  - North Western Mental Health, Melbourne, Victoria

REFERENCES:
- [Derived] Thomas N, Farhall J, Foley F, Rossell SL, Castle D, Ladd E, Meyer D, Mihalopoulos C, Leitan N, Nunan C, Frankish R, Smark T, Farnan S, McLeod B, Sterling L, Murray G, Fossey E, Brophy L, Kyrios M. Randomised controlled trial of a digitally assisted low intensity intervention to promote personal recovery in persisting psychosis: SMART-Therapy study protocol. BMC Psychiatry. 2016 Sep 7;16(1):312. doi: 10.1186/s12888-016-1024-1. PMID 27604363